CLINICAL TRIAL: NCT00674453
Title: The Effect Of Lasofoxifene On Local Mediators Of Bone Resorption In The Prevention Of Postmenopausal Osteoporosis
Brief Title: The Prevention Of Postmenopausal Osteoporosis With Lasofoxifene And Cytokine Evaluation
Acronym: LACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ligand Pharmaceuticals (Industry)
Responsible Party: Director, Project Management, Ligand Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: A2181042
Record Dates: First submitted 2008-04-30; First posted 2008-05-07 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Bone Loss
Keywords: Osteoporosis; lasofoxifene; bone density; bone markers
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — Lasofoxifene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lasofoxifene 0.25 mg/d (Experimental)
  Interventions: Drug: Lasofoxifene
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lasofoxifene — Oral tablet, 0.25 mg, daily, 2 years
  Arms: Lasofoxifene 0.25 mg/d
Other: Placebo — Matching placebo tablet given once daily for 2 years
  Arms: Placebo

SUMMARY:
The objective of the study is to demonstrate the effects that lasofoxifene has on serum markers of bone metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women over 50 years who have low bone mineral density.

Exclusion Criteria:

* Women who are under 50 years of age, are premenopausal, or who currently have osteoporosis are excluded.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2004-09; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Change in bone mineral density of the lumbar spine. | 2 years

SECONDARY OUTCOMES:
The secondary outcomes are the levels of cells and proteins in the blood that provide information about the health of bone, along with change in bone mineral density of the hip and forearm. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Sheffield, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2181042&StudyName=The%20Prevention%20Of%20Postmenopausal%20Osteoporosis%20with%20Lasofoxifene%20And%20Cytokine%20Evaluation